CLINICAL TRIAL: NCT02563743
Title: Preventing Sickness Absenteeism Among Employees With Common Mental Disorders and Stress-related Symptoms: a Cluster Randomized Trial of a Problem-solving Based Intervention Versus Care-as-usual Conducted at the Occupational Health Services
Brief Title: Stress and Mental Ill-health in the Workplace: Evaluation of an Intervention for the Prevention of Sick Leave
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gunnar Bergström, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2544/2014; 2014-0742 (Other Grant/Funding Number: Swedish Research Council for Health,Working Life and Welfare)
Record Dates: First submitted 2015-09-21; First posted 2015-09-30 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Common Mental Disorders and/or Stress Related Symptoms
Keywords: Sick-leave; Return to work; Occupational health; Common mental disorder; Depression; Anxiety disorders; Adjustment disorders; Problem solving therapy; Occupational Health Services; Randomized controlled trial; Intervention studies; Occupational stress
MeSH Terms: conditions — Depression; Anxiety Disorders; Adjustment Disorders; Occupational Stress | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Problem-solving based intervention (Experimental): Problem-solving based intervention with a participative approach. During the intervention a systematic assessment of the match between the employee and the work environment is considered. The intervention applies a participatory approach where the supervisor and the employee are guided by the OHS consultant and encouraged to actively take part in problem solving concerning the work situation. The intervention consists of three meetings, one between the OHS consultant and a representative for the employer (usually the nearest supervisor), one between the consultant and the employee and then a third meeting where all three parties participate.
  Interventions: Behavioral: Problem-solving based intervention
- Treatment as usual (Active Comparator): The control intervention consists of the usual interventions given at the participating OHS. These interventions are also work-directed and usually also include participation of both the employee and the supervisor. However, structured problem solving methods and the systematic consideration of the match between the employee and the job situation are not applied. The content of the control condition will vary between different occupational health service units.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Problem-solving based intervention — The intervention comprises both the employee and the employer, and follows a clear structure comprising problem solving, stepwise activation and relapse prevention. It includes three meetings at the OHS with additional follow-ups.
  Arms: Problem-solving based intervention
Behavioral: Treatment as usual — Study participants that are randomized into the control group will receive the usual care given at the OHS. This intervention will differ due to differences between the OHS units.
  Arms: Treatment as usual

SUMMARY:
Purpose

Common mental disorders (CMD:s) are the leading cause of sick-leave spells in Sweden, resulting in suffering for the individual and financial costs for the employer as well as for society at large. Studies on interventions that address stress and mental ill-health and that focus on sick leave and return to work (RTW) show little or no effect of commonly used methods such as medication or psychological approaches. Furthermore, these interventions often focus on the individual's symptoms without considering their work situation. The occupational health services (OHS) has knowledge of the employee's work environment and can offer treatment facilitating the employee's RTW and improving the employee's work ability while taking into account both the individual and the work situation. The intervention in the current study will be performed at the OHS.

The study aim is two-fold: first, an intervention that addresses both individual and workplace related aspects among employees with work-related CMD:s and/or stress related symptoms will be evaluated. In particular, the treatment's cost-effectiveness and impact on sick leave and mental health will be studied. Secondly, the concerned OHS staff's adherence to the intended treatment and associations with the outcome of the intervention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* The employee suffers from stress related symptoms or work-related common mental disorders.
* The employee is either not on sick leave or is on sick leave for a maximum of 3 consecutive months (full or part time).
* The employee understands both written and spoken Swedish.
* The employees nearest supervisor should be aware of the employees visit(s) at the OHS (to avoid differential selection into the experimental and the control condition)

Exclusion Criteria:

* Bullying
* Pregnancy
* Post traumatic stress-disorder
* Severe mental disorders (e.g. psychosis)
* Any co-morbidity that may substantially affect the employee's ability to work and/or quality of life.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in total registered sickness absenteeism during the 12 month follow-up period. | At baseline and 12 months after baseline.
  (1) Total sick leave in days, register data (sickness benefit and disability pension). Sickness benefit and disability pension will also be analyzed separately.
  The analyses will be repeated for outcomes on registered sick leave at a three-years follow-up

SECONDARY OUTCOMES:
Change from baseline in self-reported sickness absenteeism during the 12 months follow-up period | At baseline and during monthly follow-ups for a period of 12 months
  Self-report data obtained every four weeks during the 12-months follow-up period. These data also include short spells of sick leave.
  Possible interaction effects on the primary and secondary outcomes for (1) gender x treatment (intervention) and (2) sick leave status (sick leave/no sick leave) x treatment will be checked for and if statistically significant subgroup analyses will be considered.
The prevalence of no sick leave, part-time sick leave and full-time sick leave during the 12 months follow-up period following baseline | Twelve months after baseline
  Change from baseline in self-reported data (no sick leave, 25%, 50%, 75% or 100% sick leave) obtained every fourth week during a follow-up period of 12 months
Among those sick listed at baseline: Time to full Return to Work (RTW) during a follow-up period of 12 months | At baseline and during monthly follow-ups for a period of 12 months
  RTW will be calculated from the study inclusion date until the individual returns in ordinary hours of work during an uninterrupted period of at least four weeks. Self-reported data obtained every fourth week during a follow-up period of 12 months.
Among those sick listed at baseline: Time to Return to Work (RTW) during a follow-up period of 12 months | At baseline and during monthly follow-ups for a period of 12 months
  RTW will be calculated from the study inclusion date until the individual returns to work in any increased level (25%, 50%, 75% or 100%). Self-reported data obtained every fourth week during a follow-up period of 12 months.
Work performance impairment due to health problems | Will be assessed at baseline and once a month during a 12-month follow-up period
  Change from baseline in work performance as assessed by a question based on one item from the Work Productivity Activity Impairment - General Health Questionnaire (response format from 0-10).
Work performance impairment due to problems in working environment | Will be assessed at baseline and every other month (eighth weeks intervals) during a 12-month follow-up period
  Change from baseline in work performance as assessed by a question based on one item from the Work Productivity Activity Impairment - General Health Questionnaire (response format from 0-10).
Cost-effectiveness of the intervention compared to treatment as usual. | At 12 months after baseline
  The cost-effectiveness of the intervention will be calculated with regard to production loss (sick leave and performance while at work).
Work satisfaction | Will be assessed at baseline and after 6 and 12 months.
  Change from baseline in self-reported work satisfaction will be assessed by a single item (response format from 0-10).
Work ability index (WAI) | Will be assessed at baseline and after 6 and 12-months of study inclusion.
  Change from baseline in self-reported work ability as assessed by two items from WAI (response format from 1-5). The items relate to perceived capacity to work relative to the physical (1 item) and mental (1 item) demands of the work.
Sickness presenteeism | Will be assessed at baseline and after 6 and 12-months of study inclusion.
  Change from baseline in sickness presenteeism is assessed with a single question (response format from 1-4).
The Institute of Stress Medicine's instrument for self-rating of stress-related Exhaustion Disorder (s-ED) | Will be assessed at baseline and after 6 and 12-months of study inclusion.
  Change from baseline in self-reported exhaustion on the s-UMS (two yes/no items and one item with a response format from 0-2.
Maslach Burnout Inventory - General Survey, Exhaustion-scale | Will be assessed at baseline and after 6 and 12-months of study inclusion.
  Change from baseline in self-reported exhaustion as assessed by the MBI-GS's exhaustion scale (response format from 0 to 6).
Hospital Anxiety and Depression Scale | Will be assessed at baseline and after 6 and 12-months of study inclusion.
  Change from baseline in self-reported mental health as assessed by the Hospital Anxiety and Depression Scale (response format from 0-3).
Self-perceived health | Will be assessed at baseline and after 6 and 12-months of study inclusion.
  Change from baseline in self-perceived health will be assessed with a single question (response format from 1-5).
European Quality of Life - 5 Dimensions questionnaire (EQ-5D) | Will be measured at baseline and after 6 and 12-months of study inclusion.
  Change from baseline in self-assessed health as assessed by EQ-5D (response format from 1-3).
Self-reported stress | At baseline and every other month (eighth weeks intervals) during a follow-up period of 12 months
  Change from baseline in self-reported stress as assessed by a single item (response format from 1-5).
Karolinska Sleep Questionnaire, Insomnia sub-scale | Will be measured at baseline and after 6 and 12-months of study inclusion.
  Change from baseline in self-assessed sleeping problems as assessed by the Insomnia subscale of the Karolinska Sleep Questionnaire (response format from 1-6).
Demand-control-support model. Prognostic variable. | Baseline and at 6 and 12 months of study inclusion
  Change from Baseline at 6 and 12 months (response format from 1-4).
Other work related variables such as ongoing conflicts with the superior, perceived loss of control over work tasks and conflicts between the employee´s values and how the work actually is done. Prognostic variables. | Baseline and at 6 months after study inclusion
  Change from baseline at 6 and 12 months after baseline (Likert-type scales with 3 to 5 response options).
Physical activity. Prognostic variable. | At 6 and 12 months after intervention
  Physical activity will be assessed by a single item. Response options: 0 minutes, less than 30 minutes, 30-60 minutes, 60-90 minutes, 90-120 minutes or more than 120 minutes.
Change in work conditions. Prognostic variable. | At 6 and 12 months after intervention
  Possible changes to the participant's work conditions will be asked by a single item with 12 choices.
Change in the organization. Prognostic variable. | At 6 and 12 months after intervention
  Possible changes in the organization over the past six months are assessed with four response options.
Participants' satisfaction and experiences with the intervention or treatment as usual will be assessed at 6 months after completed intervention by eleven items (response format from 0-10 or yes/no/do not know). Process evaluation data. | Will be assessed 6 months after intervention.
  These items referred to aspects such as quality of the communication with the OHS personnel, relevance of the intervention, perceived problem-solving skills learned during the intervention, planned adjustments at work, agreement with the supervisor, the implementation of planned adjustments, if follow-up contacts with the OHS have been undertaken and questions regarding treatment satisfaction).
OHS staff's adherence to the intervention (process evaluation data) | Assessed at the end of the 12-18 months long recruitment period
  Self-reported data, single items.
Implementation of the intervention and entire research project at the OHS units (process evaluation data) | Assessed at the end of the 12-18 months long recruitment period
  Self-report data, single items and focus group interviews
Three years follow-up: Change from Baseline in registered sickness absenteeism during a 3-year follow-up period | At baseline and 3 years after baseline.
  Total sick leave in days, register data (sickness benefit and disability pension).
  The analyses will be conducted in accordance with the 12-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Bergström, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Background] Bergstrom G, Lohela-Karlsson M, Kwak L, Bodin L, Jensen I, Torgen M, Nybergh L. Preventing sickness absenteeism among employees with common mental disorders or stress-related symptoms at work: Design of a cluster randomized controlled trial of a problem-solving based intervention versus care-as-usual conducted at the Occupational Health Services. BMC Public Health. 2017 May 12;17(1):436. doi: 10.1186/s12889-017-4329-1. PMID 28494753
- [Background] Keus van de Poll M, Nybergh L, Lornudd C, Hagberg J, Bodin L, Kwak L, Jensen I, Lohela-Karlsson M, Torgen M, Bergstrom G. Preventing sickness absence among employees with common mental disorders or stress-related symptoms at work: a cluster randomised controlled trial of a problem-solving-based intervention conducted by the Occupational Health Services. Occup Environ Med. 2020 Jul;77(7):454-461. doi: 10.1136/oemed-2019-106353. Epub 2020 Apr 14. PMID 32291291
- [Background] Keus Van De Poll M, Bergstrom G, Jensen I, Nybergh L, Kwak L, Lornudd C, Lohela-Karlsson M. Cost-Effectiveness of a Problem-Solving Intervention Aimed to Prevent Sickness Absence among Employees with Common Mental Disorders or Occupational Stress. Int J Environ Res Public Health. 2020 Jul 20;17(14):5234. doi: 10.3390/ijerph17145234. PMID 32698470
- [Derived] Toropova A, Bjork Bramberg E, Bergstrom G. Return to Work Trajectories of Swedish Employees on Sick-Leave Due to Common Mental Disorders. J Occup Rehabil. 2025 Sep;35(3):479-490. doi: 10.1007/s10926-024-10216-9. Epub 2024 Jun 22. PMID 38907784